CLINICAL TRIAL: NCT04321109
Title: Alveolar Ridge Preservation Using Collagen Material and Allograft: A Randomized Controlled Trial
Brief Title: Alveolar Ridge Preservation Using Collagen Material and Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasmine Fouad (Other)
Responsible Party: Sponsor-Investigator, Yasmine Fouad, lecturer of oral medicine and periodontology, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECD 071402
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Alveolar Ridge Preservation
Keywords: Alveolar ridge preservation; Allograft; Collagen cone
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: Group (1): Seven extraction sockets that received the collagen matrix (Collacone) for alveolar ridge preservation.
  Group (2): Seven extraction sockets that were treated with mineralized cortico-cancellous bone allograft (Maxgraft) for alveolar ridge preservation
Who Masked: Outcomes Assessor
Masking Description: Results were sent to Outcome Assessor masked , so he was not able to know results belong to which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collagen cone (Experimental): Collagen matrix
  Interventions: Other: Collagen cone
- Allograft (Active Comparator): mineralized corticocancellous allograft
  Interventions: Other: Allograft

INTERVENTIONS:
Other: Allograft — Corticocancellous mineralized allograft
  Arms: Allograft
Other: Collagen cone — Collagen matrix
  Arms: Collagen cone

SUMMARY:
Seven Patients who need implants to replace non-restorable teeth in the esthetic zone.

Intervention Group (1): Seven extraction sockets that received the collagen matrix (Collagen cone) for alveolar ridge preservation.

Comparison Group (2): Seven extraction sockets that were treated with mineralized cortico-cancellous bone allograft for alveolar ridge preservation.

Outcome

1. Alveolar ridge preservation both in height and in width to improve implant success rate

   * The height of alveolar ridge was assessed clinically using a periodontal probe.
   * The width of the alveolar ridge was measured after three months after extraction using a caliper clamp.
   * Changes in the width and height of alveolar bone were evaluated in merged axial and sagittal views using the I-CAT superimposition system (CBCT).

     2- Evaluation of newly formed bone quality was performed by histological examination and histomorphometric analysis.

     3- Immuno-histochemical staining was done using polyclonal antibody to detect (BMP-2) marker of bone formation

DETAILED DESCRIPTION:
The aim of the present study was to compare three months post-extraction augmented ridge using collagen matrix versus mineralized cortico-cancellous bone allograft. This comparison was done clinically, histologically, immunohisto-chemically and radiologically.

• Clinical parameters included; vertical bone height and bone width that were recorded at baseline and at three months after extraction. Moreover, histomorphometric parameters included; area fraction of osteoid and mature bone three months after extraction by histomorphometric analysis. Immunohistochemical analysis using polyclonal antibody to detect BMP-2 marker of bone formation. Radiographic parameters included superimposition of baseline CBCT, three months after extraction and another one six months after loading with subsequent measurement of bone height, bone width and bone density.

A core biopsy was taken three months after tooth extraction which has undergone histomorphometric and immunohistochemical analysis; implant placement was also done at the same time.

In the present study, it was found that the mean bone height decreased with a higher percent in collagen matrix group than mineralized cortico-cancellous bone allograft group with a non significant difference between both groups.

In addition, this study showed that the mean bone width decreased more in collagen matrix group than mineralized cortico-cancellous bone allograft group with a non significant difference between them.

Moreover, in the present study, Histomorphometric analysis revealed new bone trabeculae formation with osteoblastic rimming, the surrounding fibrous tissue is cellular and remnants of the graft materials was detected , with no marked difference in the amount of newly formed bone between two groups .

Regarding immunohistochemical analysis in both groups, the osteoblasts in the fibrous tissue and osteocytes in newly formed bone are showing nuclear staining, with increasing area of immunopositive cells in mineralized cortico-cancellous bone allograft group.

Radiographically, CBCT superimposition revealed that a greater percent decrease in bone height was denoted in collagen matrix than mineralized cortico-cancellous bone allograft group with a significant difference between both groups after 3 and 6 months.

Accordingly bone width showed a higher decrease in mineralized cortico-cancellous bone allograft group than Collagen matrix group with a non significant difference between both groups after 3 and 6 months.

Finally, bone density showed a greater decrease in Collagen matrix group than mineralized cortico-cancellous bone allograft group with a non significant difference after 3 months but significant difference was found after 6 months between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were medically free .
2. Two teeth indicated for extraction due to either severe decay, tooth fracture or failed endodontic treatment.

Exclusion Criteria:

1. Patients with poor oral hygiene or not willing to perform oral hygiene measures.
2. Pregnant and breast-feeding females.
3. Smokers , Teeth with periodontal or periapical infections.
4. Patients with malocclusion.
5. All patients who had known contraindication to dental implant surgery (e.g: bleeding tendency, radiotherapy, taking bisphosphonate)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
clinical score | change from baseline at 12 weeks
  Dimensional changes in alveolar ridge after alveolar ridge preservation both clinically and radiographically

SECONDARY OUTCOMES:
BMP-2 | detected at 12 weeks
  Bone morphogenic protein -2 immunopositive cells in immunostained sections

CONTACTS AND LOCATIONS:
Overall Officials: Hala A Abuel-Ela, Professor, Study Director — Faculty of Dentistry Ain Shams University